CLINICAL TRIAL: NCT01536366
Title: Effect of BIA 9-1067 on the Pharmacokinetics of Repaglinide in Healthy Volunteers
Brief Title: Effect of BIA 9-1067 on the Pharmacokinetics of Repaglinide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-115
Record Dates: First submitted 2012-01-23; First posted 2012-02-22 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Period 1: BIA 9-1067 + repaglinide Period 2: Repaglinide
  Interventions: Drug: BIA 9-1067; Drug: Repaglinide
- Group 2 (Experimental): Period 1: Repaglinide Period 2: BIA 9-1067 + repaglinide
  Interventions: Drug: BIA 9-1067; Drug: Repaglinide

INTERVENTIONS:
Drug: BIA 9-1067 — 25 mg BIA 9-1067 (single-dose)
  Other Names: OPC, Opicapone
Drug: Repaglinide — 0.5 mg repaglinide (single-dose)
  Other Names: Novonorm®

SUMMARY:
The purpose of this study is to investigate the CYP2C8 inhibition by BIA 9-1067.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, two-way crossover study in healthy young male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or ex-smokers for at least 3 months.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* Any abnormality in the coagulation tests.
* Any abnormality in the liver function tests.
* A history of relevant atopy or drug hypersensitivity.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to each treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Had used medicines within 2 weeks of admission to first period that may have affected the safety or other study assessments, in the investigator's opinion.
* Had previously received BIA 9-1067.
* Had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Had participated in more than 2 clinical trials within the 12 months prior to screening.
* Had donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or had medical dietary restrictions.
* Cannot communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to gave written informed consent.
* Employees at BIAL - Portela & Cª, S.A.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not used an approved effective contraceptive method (double-barrier or intra-uterine device) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, MD, PhD, Principal Investigator — BIAL - Portela & Cª S.A.
Locations (1):
- Bial - Portela & Cª, S.A., S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 14 | 13
BIA 9-1067 + Repaglinide | 14 | 10
Repaglinide | 14 | 13
Follow-up | 13 | 9
Completed | 1 | 9
Not Completed | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 + Repaglinide: BIA 9-1067 25 mg Repaglinide 0.5 mg
- Repaglinide: Repaglinide 0.5 mg
Arm/Group | BIA 9-1067 + Repaglinide | Repaglinide
Number analyzed (Participants) | 24 | 27
ng/mL
  BIA 9-1067 | 400 (245.2) | NA (NA) — BIA 9-1067 was not administered.
  Repaglinide | 11.6 (5.22) | 9.76 (5.42)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose.
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 + Repaglinide | Repaglinide
Number analyzed (Participants) | 24 | 27
hours
  BIA 9-1067 | 2.00 [1.0 to 4.0] | NA [NA to NA] — BIA 9-1067 was not administered
  Repaglinide | 0.5 [0.5 to 0.75] | 0.50 [0.5 to 3.0]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 + Repaglinide | Repaglinide
Number analyzed (Participants) | 24 | 27
ng.h/mL
  BIA 9-1067 | 979 (607) | NA (NA) — BIA 9-1067 was not administered
  Repaglinide | 14.2 (4.96) | 13.1 (5.33)

4. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve From Time 0 to Infinity
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 + Repaglinide | Repaglinide
Number analyzed (Participants) | 24 | 27
ng.h/mL
  BIA 9-1067 | 1015 (608) | NA (NA) — BIA 9-1067 was not administered
  Repaglinide | 15.0 (4.95) | 14.1 (5.5)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 + Repaglinide | Repaglinide
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 7/24 | 8/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 + Repaglinide (N=24) | Repaglinide (N=27)
Presyncope (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes